CLINICAL TRIAL: NCT02188368
Title: A Phase 2 Study of Pomalidomide as a Replacement for Lenalidomide for Multiple Myeloma Patients Relapsed or Refractory to a Lenalidomide-Containing Combination Regimen
Brief Title: Pomalidomide for Lenalidomide for Relapsed or Refractory Multiple Myeloma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Oncotherapeutics (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PO-CL-MM-PI-003854
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
Keywords: Pomalidomide; Lenalidomide refractory; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Steroids; Dexamethasone; Prednisone; 1-dodecylpyridoxal; carfilzomib; Bortezomib; Clarithromycin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: POM 4mg+Steroids+(CFZ, BTZ, CY or CLA) (Experimental): POM 4 mg PO days 1-21 Steroids at the same dose and on the same days as the patient's lenalidomide-containing treatment (it varies for each subject).
  BTZ (bortezomib) at the same dose and on the same days as the patient's lenalidomide-containing treatment (it varies for each subject).
  CFZ (carfilzomib) at the same dose and on the same days as the patient's lenalidomide-containing treatment (it varies for each subject).
  CLA (clarithromycin) at the same dose and on the same days as the patient's lenalidomide-containing treatment (it varies for each subject).
  CY (cyclophosphamide) at the same dose and on the same days as the patient's lenalidomide-containing treatment (it varies for each subject).
  Interventions: Drug: POM; Drug: Steroids; Drug: CFZ; Drug: BTZ; Drug: CLA; Drug: CY
- B: POM 3mg+PLD with or without steroids (Experimental): POM 3 mg PO days 1-21 Steroids (if the patient had received them) at the same dose and on the same days as the patient's lenalidomide-containing treatment (it varies for each subject).
  PLD at the same dose and on the same days as the patient's lenalidomide-containing treatment (it varies for each subject).
  Interventions: Drug: POM; Drug: Steroids; Drug: PLD
- C: POM MTD + other drugs (Experimental): Phase 1:
  POM at escalating doses of 2 mg (Cycle 1), 3 mg (Cycle 2) or 4 mg (Cycle 3+) All other agents at the same dose and on the same days as the patients were receiving them in the lenalidomide-containing regimen they had failed
  Phase 2:
  POM at the MTD All other agents, at the same dose and on the same days as phase 1
  Interventions: Drug: POM

INTERVENTIONS:
Drug: POM
  Other Names: Pomalidomide; Pomalyst; Actimid; CC-4047
Drug: Steroids
  Other Names: Dexamethasone; prednisone; methyprednisolone
  Arms: A: POM 4mg+Steroids+(CFZ, BTZ, CY or CLA); B: POM 3mg+PLD with or without steroids
Drug: PLD
  Other Names: Pegylated liposomal doxirrubicin
  Arms: B: POM 3mg+PLD with or without steroids
Drug: CFZ
  Other Names: Carfilzomib; Kyprolis
  Arms: A: POM 4mg+Steroids+(CFZ, BTZ, CY or CLA)
Drug: BTZ
  Other Names: Bortezomib; Velcade
  Arms: A: POM 4mg+Steroids+(CFZ, BTZ, CY or CLA)
Drug: CLA
  Other Names: Clarithromycin
  Arms: A: POM 4mg+Steroids+(CFZ, BTZ, CY or CLA)
Drug: CY
  Other Names: Cyclophosphamide
  Arms: A: POM 4mg+Steroids+(CFZ, BTZ, CY or CLA)

SUMMARY:
The purpose of this clinical research study is to evaluate the safety and effectiveness (good and bad effects) of pomalidomide given as part of a combination therapy that include more than just steroids to treat subjects with relapsed (subjects whose disease came back) or refractory (subjects whose disease did not respond to past treatment) multiple myeloma (MM).

Pomalidomide (alone or in combination with dexamethasone) has been approved by the United States Food and Drug Administration (FDA) for the treatment of MM patients who have received at least two prior therapies, including lenalidomide and bortezomib, and have demonstrated disease progression on or within 60 days of completion of their last therapy. However, the use of pomalidomide in combination with other drugs used to treat MM, such as chemotherapeutic agents and proteasome inhibitors, is currently being tested and is not approved. Pomalidomide is in the same drug class as thalidomide and lenalidomide. Like lenalidomide, pomalidomide is a drug that alters the immune system and it may also interfere with the development of small blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells. The testing done with pomalidomide thus far has shown that it is well-tolerated and effective for subjects with MM both on its own and in combination with dexamethasone. Using another drug class, namely proteasome inhibitors, we have demonstrated that simply replacing a proteasome inhibitor with another in an established anti-myeloma treatment regimen can frequently overcome resistance regardless of the other agents that are part of the anti-myeloma regimen. Importantly, the toxicity profile of the new combinations closely resembled that of the proteasome inhibitor administered as a single agent. Based on this experience, we hypothesize that the replacement of lenalidomide with pomalidomide will yield similar results in a similar relapsed/refractory MM patient population.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, open-label and non-randomized study to evaluate the efficacy and safety of pomalidomide as a replacement for lenalidomide among MM patients who have failed lenalidomide-containing regimens that include more than steroids within 6 months of their last dose of lenalidomide. Pomalidomide will replace lenalidomide in a combination regimen containing an alkylating agent (cyclophosphamide), anthracycline (doxorubicin or PLD), proteasome inhibitor (bortezomib or carfilzomib) and/or a glucocorticosteroid (prednisone, dexamethasone or methylprednisolone). Pomalidomide will be administered on days 1-21 of a 28-day cycle, whereas other drugs (anthracyclines, proteasome inhibitors, steroids or alkylating agents except melphalan) will be administered using the same schedule(s), dose(s) and drug combination as the last lenalidomide-containing regimen that the patient received and failed. This study will enroll patients resistant to a lenalidomide-containing combination regimen as demonstrated by PD while being treated or that has relapsed within 6 months of the last dose of lenalidomide in their last lenalidomide-containing combination regimen or while on lenalidomide or lenalidomide and steroid maintenance therapy. Forty-five patients will be enrolled in the study.

The study consists of: 1) a screening period; 2) up to eight 28-day, treatment cycles; 3) a final assessment to occur 28 days after the end of the last treatment cycle; and 4) a follow-up period.

Subjects eligible for this study will receive treatment with study drug for a maximum of eight 28-day treatment cycles, depending on the schedule of their last lenalidomide-containing regimen. Subjects are to be treated to a maximum response (lowest level of paraprotein) plus 1 additional cycle, without exceeding a total of 8 cycles, or complete 8 cycles of therapy without progressing (PD).

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a diagnosis of MM based on standard criteria as follows:

   * Major criteria:

     1. plasmacytomas on tissue biopsy
     2. bone marrow plasmacytosis (greater than 30% plasma cells)
     3. monoclonal immunoglobulin (Ig) spike on serum electrophoresis IgG greater than 3.5 g/dL or IgA greater than 2.0 g/dL; kappa or lambda light chain excretion greater than 1 g/day on 24-hour urine protein electrophoresis
   * Minor criteria:

     1. bone marrow plasmacytosis (10% to 30% plasma cells)
     2. monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
     3. lytic bone lesions
     4. normal IgM less than 50 mg/dL, IgA less than 100 mg/dL, or IgG less than 600 mg/dL
   * Any of the following sets of criteria will confirm the diagnosis of multiple myeloma:

     * any 2 of the major criteria
     * major criterion 1 plus minor criterion 2, 3, or 4
     * major criterion 3 plus minor criterion 1 or 3
     * minor criteria 1, 2, and 3, or 1, 2, and 4
2. Currently has progressive MM that has relapsed while currently receiving or within 6 months of receiving the maximum tolerated dose of lenalidomide at the physician's discretion as part of a combination treatment that includes more than just steroids in a 21-day or a 28-day cycle schedule. MM patients that are relapsed or have refractory disease, as defined below, are both eligible for enrollment provided they fulfill the other eligibility criteria:

   * Patients are refractory to a lenalidomide combination regimen, when they progress while currently receiving the lenalidomide combination treatment or within 8 weeks of its last dose.
   * Patients are considered relapsed, when they progress between 8 and 26- weeks from their last dose of lenalidomide as part of a lenalidomide-combination therapy that includes more than just steroids.
   * Prior treatment with four days or less of a total of 400 mg of prednisone (or an equivalent potency of another steroid) for MM will not be considered a regimen
3. Currently has MM with measurable disease, defined as:

   * a monoclonal immunoglobulin spike on serum electrophoresis of at least 0.5 g/dL and/or
   * urine monoclonal protein levels of at least 200 mg/24 hours
   * for patients without measurable serum and urine M-protein levels, an abnormal free light chain ratio (normal value: 0.26 - 1.65)
   * Serum free light chain (SFLC) > 100 mg/L (involved light chain) and abnormal ƙ/λ ratio
4. Patients with previous clotting or thrombotic events must be able to take aspirin (acetylsalicylic acid, ASA) at 81 or 325 mg /daily as prophylactic anticoagulation (subjects intolerant to ASA may use warfarin or low molecular weight heparin) and/or antithrombotic agents.

Key Exclusion Criteria:

1. Plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes (POEMS) syndrome
2. Plasma cell leukemia
3. Primary amyloidosis
4. Non-hematologic malignancy within the past 5 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
5. Impaired cardiac function or clinically significant cardiac diseases, including myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class II or greater heart failure, uncontrolled angina, clinically significant pericardial disease, severe uncontrolled ventricular arrhythmias, echocardiogram or multigated acquisition scan (MUGA) evidence of left ventricular ejection fraction (LVEF) below institutional normal within 28 days prior to enrollment, electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
6. Received the following prior therapy:

   * Pomalidomide
   * Lenalidomide alone or in combination with steroids in their last treatment regimen. Interim therapy not containing lenalidomide between their last lenalidomide-containing regimen and the start of the trial.
   * A melphalan-containing regimen as the immediate prior line of treatment
   * Chemotherapy within 3 weeks of study drugs (6 weeks for nitrosoureas)
   * Corticosteroids (>10 mg /daily prednisone or equivalent) within 3 weeks of study drugs
   * Immunotherapy or antibody therapy as well as thalidomide, lenalidomide, arsenic trioxide or bortezomib within 21 days before study drugs
   * Extensive radiation therapy within 28 days before study drugs. Receipt of localized radiation therapy does not preclude enrollment.
   * Use of any other experimental drug or therapy within 28 days of study drugs
7. Known hypersensitivity to compounds of similar chemical or biological composition to thalidomide and lenalidomide.
8. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Cycles 1-3 for selected regimens (up to 3 months)
  MTD will be determined for any ≥ three-drug combinations other than:
  bortezomib + steroids + lenalidomide; carfilzomib + steroids + lenalidomide; clarithromycin + steroids + lenalidomide; cyclophosphamide + steroids + lenalidomide pegylated liposomal doxorubicin (PLD) + lenalidomide with or without steroids
Number of subjects with adverse events | up to 36 months
  Adverse events will be graded via the Common Terminology Criteria for Adverse Events (CTCAE) v 4.03 criteria.
Overall Response Rate | up to 36 months
  Overall response rate (ORR): complete response (CR)+ very good partial response (VGPR) + partial response (PR)
Clinical Benefit Rate (CBR) | up to 36 months
  CBR=ORR + minor response (MR)

SECONDARY OUTCOMES:
Time to Progression | time from initiation of therapy to progressive disease (assessed at least over 36 months)
  The time from the initiation of therapy to progressive disease
Progression-free survival (PFS) | time from initiation of therapy to progressive disease or death from any cause, whichever comes first (assessed at least over 36 months)
  Time from initiation of therapy to progressive disease or death from any cause, whichever occurs first
Time to first response (TTP) | time from initiation of therapy to the first evidence of a confirmed response (up to 36 months)
  time from initiation of therapy to the first evidence of a confirmed response
Duration of response (DOR) | time from the first response (> PR) to progressive disease (assessed at least over 36 months)
  time from the first response (> PR) to progressive disease
Overall survival (OS) | time from initiation of therapy to death from any cause or last follow-up visit (assessed at least over 36 months).
  time from initiation of therapy to death from any cause or last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: James R Berenson, MD, Principal Investigator — James R. Berenson MD, Inc.
Locations (12):
- United States (12):
  - California Cancer Associates for Research & Excellence (cCARE), Encinitas, California
  - Compassionate Care Research Group, Fountain Valley, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - Inland Hematology Oncology Medical Group, Inc, San Bernardino, California
  - Wellness Oncology and Hematology, West Hills, California
  - James R. Berenson, MD, Inc., West Hollywood, California
  - VA Sierra Nevada, Reno, Nevada
  - San Juan Oncology Associates, Farmington, New Mexico
  - Gabrail Cancer Center, Canton, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Wellmont Medical Associates Oncology and Hematology, Kingsport, Tennessee
  - Vista Oncology, Olympia, Washington